CLINICAL TRIAL: NCT01502501
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Cardiovascular Effects of Intramyocardial and Intravenous Implantation of Autologous Adipose-Derived Stem Cells in Non-Ischemic Congestive Heart Failure Patients
Brief Title: Safety and Efficacy of Adipose Derived Stem Cells for Non-Ischemic Congestive Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-CHF-001
Record Dates: First submitted 2011-12-27; First posted 2011-12-30 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Non-Ischemic Congestive Heart Failure
Keywords: CHF; Heart Failure; Non-Ischemic; nonischemic; nonischemia
MeSH Terms: conditions — Heart Failure | interventions — HMGA2 Protein; Lipectomy; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Harvesting and Implantation of Adipose-Derived Stem Cells (ASCs) — Local liposuction procedure to harvest the fat tissue. Adipose Derived Stem Cells are then implanted via intramyocardial and intravenous injection.
  Other Names: Lipo; Liposuction; Catheter; IV; ADSC

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with Heart Disease as assessed by a series of measurements indicating improvement, stability, or degradation of a patient's cardiovascular function and exercise capacity?

DETAILED DESCRIPTION:
This will be an open-label, non-randomized, multi-center patient-sponsored study designed to assess the safety and cardiovascular effects of Adipose-derived Stem Cell (ASC) implantation using a catheter delivery system in patients who have nonischemic congestive heart failure. A percutaneous transluminal endomyocardial injection catheter will be used for delivery of ASCs. The therapy is composed of cells isolated from a patient's own adipose tissue. Liposuction will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent
2. Age >18 years and < 80 years
3. NYHA Class II-IV
4. Congestive Heart Failure without an acute coronary syndrome during the prior 6 months
5. LVEF less than or equal to 40% measured by echocardiography at both local and investigative sites, AND

   * Left ventricular wall without mural thrombus and of thickness greater than 0.5 cm
   * No significant valvular disease including: Moderate-to-severe mitral regurgitation (3-4+), aorticstenosis (valve area <1.5 cm2), aortic insufficiency (3-4+)
6. Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

1. Limiting symptoms due to non-CHF causes, such as lung disease, peripheral vascular disease, arthritis or other musculoskeletal disorders
2. Inability to complete a 6-minute walk test for any reason
3. Need for intravenous CHF medications, chronic continuous oxygen therapy or oral steroids,
4. Coronary Artery Bypass Surgery (CABG) surgery within 60 days prior to screening
5. Planned revascularization within 4 months following enrollment
6. Aortic aneurysm or dilatation (>3.8 cm by echocardiography or other imaging modality)
7. Peripheral vascular disease at or below the distal aorta that may interfere with catheter use
8. Hemodynamically significant pericardial disease
9. Prior aortic or mitral valve replacement
10. Biventricular pacing device implant within the last 3 months OR whose device is scheduled to be revised following enrollment in this trial
11. Scheduled to receive or history of cardiac transplant, surgical remodeling procedure, left ventricular assist device
12. Stroke within 180 days of screening
13. Positive pregnancy test in women of child bearing potential or who are unwilling to use an acceptable method of contraception.
14. Drug or alcohol dependence
15. Life expectancy of less than 1 year
16. History of cancer (other than non-melanoma skin cancer or in situ cervical cancer) in the last five years
17. Exposure to angiogenic therapy (including myocardial laser) or another investigational drug within 60 days of screening, or enrollment in any concurrent study that may confound the results of this study
18. Any factors in the opinion of the Investigator which render the patient unsuitable for participation, that will interfere with conduct of the study or interpretation of the results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in 6 minute walk test | 3 months
  compared to baseline
Minnesota Living with Heart Failure Quality of Life Questionnaire | 3 months
Improvement in 6 minute walk test | 6 months
Minnesota Living with Heart Failure Quality of Life Questionnaire | 6 months
Number of Adverse Events | 6 months

SECONDARY OUTCOMES:
Improvement in New York Heart Association (NYHA) classification | 3 months
Improvement in the Left Ventricular Ejection Fraction (LVEF) | 3 months
  Determined by and echo
Improvement in the Left Ventricular (LV) Volume | 3 months
  Determined by an echo
Improvement in New York Heart Association (NYHA) classification | 6 months
Improvement in the Left Ventricular Ejection Fraction (LVEF) | 6 months
Improvement in the Left Ventricular (LV) Volume | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Parcero, MD, Principal Investigator — Instituto de Medicina Regenerativa
Locations (1):
- Instituto de Medicina Regenerativa, Tijuana, Estado de Baja California, Mexico